CLINICAL TRIAL: NCT03094923
Title: Effects of Preoperative Inspiratory Muscle Training on Functional Capacity and Pulmonary Complications in Coronary Artery Bypass Graft Surgery
Brief Title: Effects of Respiratory Muscle Training on Postoperative Pulmonary Complications of Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Kelly Cattelan Bonorino, Post graduation, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1632008
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Heart Diseases; Coronary Disease; Cardiovascular Diseases; Coronary Artery Occlusion
MeSH Terms: conditions — Heart Diseases; Coronary Disease; Cardiovascular Diseases; Coronary Occlusion | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): Inspiratory muscle training with threshold device and workloud 30% of the peak inpiratory preassure, during two weeks prior to surgery, seven days a week, twice a day, three sets of ten repetitions with supervision.
  Interventions: Other: Inspiratory Muscle Training
- Control group (No Intervention): Control group will receive a supportive educational component in the preoperative period.

INTERVENTIONS:
Other: Inspiratory Muscle Training — The inspiratory muscle training (IMT) will be carried out in the IG with Threshold® IMT (Respironics New Jersey, Inc) consisting of a unidirectional flow control valve which assures the constant resistance (linear load) between 7 and 41cmH20.
  The IMT will be carried out in the sitting position with a load of 30% of the MIP during the two weeks preceding the surgery, seven days a week, twice daily in three series of ten repetitions with a 30 second interval between series, under the supervision of a physiotherapist. A load of 15% of the MIP was used only on the first day of training in order for the individual to adapt to the equipment. Subsequently, the 30% MIP load will be applied and readjusted according to the new MIP values determined every four days.
  Other Names: Respiratory Muscle Training
  Arms: Inspiratory muscle training

SUMMARY:
This study will evaluate the profilatic effects of inspiratory muscle training (IMT) on functional capacity, respiratory muscle strength, postoperative pulmonary complications and days of hospitalization (PPC) in patients submitted to coronary artery bypass graft surgery (CABG).

DETAILED DESCRIPTION:
Patients undergoing coronary artery bypass graft surgery are at risk of postoperative pulmonary complications, which lead to increased postoperative morbidity and mortality.

A few studies have demonstrated that preoperative physical therapy has advantages over postoperative care in patients undergoing cardiac . In this way, this study aim to investigate the effects of preoperativeinspiratory muscle training in patients at high risk of postoperative pulmonary complications who were scheduled for coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* High-risk patients underwent primary elective CABG (Coronary artery bypass graft), High-risk will be defined as 2 or more the following: age>70 years; cough and expectoration; diabetes; smoker; COPD (Chronic Obstructive Pulmonary Disease)

Exclusion Criteria:

* Uncontrolled arrhythmia,
* Decompensated heart failure,
* Unstable angina upon selection or during the inspiratory muscle training (IMT),
* Need for reoperation and association of another procedure during surgery (e.g. valve correction associated with CABG)
* Severe orthopedic or neurological conditions.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01-12 (Actual); Primary Completion 2011-03-17 (Actual); Study Completion 2014-01-18 (Actual)

PRIMARY OUTCOMES:
Postoperative Pulmonary Complications | 1 month
  The postoperative pulmonary complications (PPC) will be classified according to an ordinal scale from 1 to 4 , as proposed by Kroenke (2002).
  The PPCs will be defined as clinically significant if the individual presented two or more Level 2 items or one or more Level 3 and/or 4 items. The Level 1 items were considered subclinical.

SECONDARY OUTCOMES:
Respiratory Muscle Strenght | 1 month
  The respiratory muscle strength will be determined by means of a calibrated analogical manovacuometer, graded from -120 to +120cmH20, defining the maximum inspiratory and expiratory pressure (MIP and MEP). The MEP will be measured by the patient's maximum inflation of the lungs (total lung capacity), followed by a maximum forced expiration lasting 1 second. The maximum inspirator pressure (MIP) assessment will be carried out by the patient's maximum expiration, followed by a maximum inspiratory force lasting 1 second. At least three technically acceptable measurements will be carried out, presenting a difference of 10% or less among the values. The analysis considered the highest value (Neder, 1999; Hulzebous, 2006)
Functional Capacity | 1 month
  The functional capacity will be assessed by means of a 6-minute walk test (T6min) in accordance with the "American Thoracic Society - ATS" guidelines. Two tests will carried out, with a thirty minute interval between them, at a flat location inside the hospital. The 30 meter distance to be covered in a straight line will be marked with a measuring tape. The patient's performance will be assessed according to the longest distance covered (Holland et al, 2014)
Lenght of hospital stay hospitalization | 1 month
  The postoperative length of stay in hospital will be assessed by calculating the number of days the patient in the hospital from the day of the surgery until the hospital discharge authorized by the cardiology team physician.

IPD SHARING:
Plan to Share IPD: No